CLINICAL TRIAL: NCT06663566
Title: Application of FAPI Visualization in the Assessment of Right Ventricular Dysfunction Due to Volume Overload
Status: Enrolling by invitation | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xiaozheng Zhou, Doctor, Department of Cardiovascular Surgery, Beijing Anzhen Hospital, Capital Medical University, Beijing Institute of Heart, Lung and Vessel Disease, Beijing 100029, China, Beijing Anzhen Hospital
Other Study IDs: KS2024071
Record Dates: First submitted 2024-10-23; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Right Heart Insufficiency; Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- high-FAPI+: FAPI Nuclear Medicine Cardiac Imaging stronge Positive" in English.
  Interventions: Diagnostic Test: Diagnose the patient's right heart function as well as right heart fibrosis
- low-FAPI+: FAPI Nuclear Medicine Cardiac Imaging Weak Positive" in English.
  Interventions: Diagnostic Test: Diagnose the patient's right heart function as well as right heart fibrosis
- No FAPI+: FAPI nuclear medicine cardiac imaging negative
  Interventions: Other: Diagnose the patients right heart function as well as right heart fibrosis

INTERVENTIONS:
Other: Diagnose the patients right heart function as well as right heart fibrosis — Diagnose the patients right heart function as well as right heart fibrosis
  Groups: No FAPI+
Diagnostic Test: Diagnose the patient's right heart function as well as right heart fibrosis — Diagnose the patient's right heart function as well as right heart fibrosis
  Groups: high-FAPI+
Diagnostic Test: Diagnose the patient's right heart function as well as right heart fibrosis — Diagnose the patient's right heart function as well as right heart fibrosis
  Groups: low-FAPI+

SUMMARY:
"Bicuspid aortic stenosis represents the most prevalent form of cardiac valve disease, primarily resulting from degenerative alterations and rheumatic conditions that disrupt mitral valve function. This dysfunction exacerbates the hemodynamic burden on the right heart, leading to secondary pulmonary hypertension-a condition uniquely predisposed to myocardial fibrosis. The role of right ventricular (RV) fibrosis in pulmonary hypertension induced by bicuspid aortic stenosis remains an area of active investigation. Modifications in the extracellular matrix collagen network may mitigate excessive dilation of the pressure-overloaded right ventricle; however, fibrosis concurrently compromises cardiac performance. An increasing body of experimental evidence indicates that fibrosis is pivotal in both the onset and progression of right ventricular dysfunction. In cases of secondary pulmonary hypertension, the right ventricle endures a posterior load approximately five times greater than normal, rendering these circumstances an excellent model for examining pressure loading effects on RV structure. Notably, severe RV fibrosis persists even after hemodynamic normalization following mitral valve repair; thus, preoperative evaluation of RV fibrosis is essential for optimizing patient outcomes in individuals with secondary pulmonary hypertension attributable to bicuspid aortic stenosis.

In recent years, myocardial nuclear imaging has gained prominence as a tool for assessing myocardial fibrosis. Initial studies investigated FAPI myocardial nuclear imaging's efficacy in evaluating left ventricular fibrosis among patients with aortic stenosis; subsequent research elucidated its correlation with sudden cardiac death risk in individuals suffering from obstructive hypertrophic cardiomyopathy.

The comprehension regarding how myocardial fibrosis impacts right ventricular function within patients experiencing pulmonary hypertension due to bicuspid aortic stenosis remains limited. The association between histological RV fibrosis and adverse prognostic indicators as well as outcomes related to right heart failure warrants further exploration."

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Tricuspid valve insufficiency; must understand the purpose of the study and signed an informed consent form;

Exclusion Criteria:

Combined coronary artery stenosis; Combined with aortic aneurysm related diseases; Patients with congenital heart disease;

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study was performed in patients with volumetric right ventricular dysfunction. To evaluate the right ventricular function in patients with valvular heart disease and optimize the condition detection and volume therapy in patients with right ventricular dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Right heart dysfunction | 15 days
  Central venous pressure（cmH2O）
Right heart dysfunction | 3 mouths
  P-V Curve of curve（cmH2O）
Right heart dysfunction | 15 days
  Duration of tracheal intubation（d)
Right heart dysfunction | 15 days
  P-V Curve of curve
Right heart dysfunction | 15 days
  TAPSE
Right heart dysfunction | 3 mouths
  TAPSE

CONTACTS AND LOCATIONS:
Locations (1):
- FAPI, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ye Y, Desai R, Vargas Abello LM, Rajeswaran J, Klein AL, Blackstone EH, Pettersson GB. Effects of right ventricular morphology and function on outcomes of patients with degenerative mitral valve disease. J Thorac Cardiovasc Surg. 2014 Nov;148(5):2012-2020.e8. doi: 10.1016/j.jtcvs.2014.02.082. Epub 2014 Mar 1. PMID 24698557
- [Result] Le Tourneau T, Deswarte G, Lamblin N, Foucher-Hossein C, Fayad G, Richardson M, Polge AS, Vannesson C, Topilsky Y, Juthier F, Trochu JN, Enriquez-Sarano M, Bauters C. Right ventricular systolic function in organic mitral regurgitation: impact of biventricular impairment. Circulation. 2013 Apr 16;127(15):1597-608. doi: 10.1161/CIRCULATIONAHA.112.000999. Epub 2013 Mar 13. PMID 23487435
- [Result] Towheed A, Sabbagh E, Gupta R, Assiri S, Chowdhury MA, Moukarbel GV, Khuder SA, Schwann TA, Bonnell MR, Cooper CJ, Khouri S. Right Ventricular Dysfunction and Short-Term Outcomes Following Left-Sided Valvular Surgery: An Echocardiographic Study. J Am Heart Assoc. 2021 Feb 16;10(4):e016283. doi: 10.1161/JAHA.120.016283. Epub 2021 Feb 9. PMID 33559474
- [Result] Purmah Y, Lei LY, Dykstra S, Mikami Y, Cornhill A, Satriano A, Flewitt J, Rivest S, Sandonato R, Seib M, Lydell CP, Howarth AG, Heydari B, Merchant N, Bristow M, Fine N, Gaztanaga J, White JA. Right Ventricular Ejection Fraction for the Prediction of Major Adverse Cardiovascular and Heart Failure-Related Events: A Cardiac MRI Based Study of 7131 Patients With Known or Suspected Cardiovascular Disease. Circ Cardiovasc Imaging. 2021 Mar;14(3):e011337. doi: 10.1161/CIRCIMAGING.120.011337. Epub 2021 Mar 16. PMID 33722059
- [Result] Kresoja KP, Rommel KP, Lucke C, Unterhuber M, Besler C, von Roeder M, Schober AR, Noack T, Gutberlet M, Thiele H, Lurz P. Right Ventricular Contraction Patterns in Patients Undergoing Transcatheter Tricuspid Valve Repair for Severe Tricuspid Regurgitation. JACC Cardiovasc Interv. 2021 Jul 26;14(14):1551-1561. doi: 10.1016/j.jcin.2021.05.005. PMID 34294396